CLINICAL TRIAL: NCT02545647
Title: Banded Versus Non-banded Roux-en-y Gastric Bypass, a Randomised Controlled Trial
Brief Title: Banded Versus Non-banded Roux-en-y Gastric Bypass
Acronym: Bandolera
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0624
Record Dates: First submitted 2015-09-03; First posted 2015-09-10 (Estimated); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard RYGB (No Intervention): 65 patients undergo a standard Roux-en-Y gastric bypass
- Banded RYGB (Active Comparator): 65 patients undergo a banded RYGB (BRYGB)
  Interventions: Device: BRYGB

INTERVENTIONS:
Device: BRYGB — 65 patients undergo a banded RYGB
  Other Names: banded RYGB
  Arms: Banded RYGB

SUMMARY:
A Roux-en-Y Gastric Bypass (RYGB) is on the long term not always successful in every patient because weight regain can occur. An intervention to prevent weight regain in the future is to place a silicone band (non-adjustable) around the pouch of the RYGB (Banded-RYGB: BRYGB) which increases weight loss and decreases weight regain on the longer term. The question is whether primary application of a banded bypass gives a greater weight loss and / or prevent weight regain in the future versus a standard RYGB.

DETAILED DESCRIPTION:
A Roux-en-Y Gastric Bypass (RYGB) is on the long term not always successful in every patient because weight regain can occur. An intervention to prevent weight regain in the future is to place a silicone band (non-adjustable) around the pouch of the RYGB (Banded-RYGB: BRYGB) which increases weight loss and decreases weight regain on the longer term. The question is whether primary application of a banded bypass gives a greater weight loss and / or prevent weight regain in the future versus a standard RYGB.

The Study design is a prospective, randomized, single center study.

Study population: patients who qualify for a RYGB are eligible to participate. The primary RYGB patients may participate if there is a BMI of 35 kg / m2 with a morbidly obesity-related comorbidity or a BMI of 40kg / m2 or higher.

Intervention: The standard RYGB with a vertical pouch over a 40 french feeding tube with a volume of 30-50 ml, is compared with a banded-RYGB (BRYGB)

ELIGIBILITY:
Inclusion Criteria:

* all patients who are eligible for a primary RYGB

Exclusion Criteria:

* Bariatric surgery in history
* Patients with a language barrier which may affect the compliance with medical advice
* Any kind of genetic disorders which can be of influence on the monitoring of medical advice
* Patients with a disease not related to morbid obesity, such as Cushing or drug related.
* Chronic bowel disease for example Crohn's disease or colitis Colitis.
* Renal impairment (MDRD <30) or hepatic dysfunction (liver function twice the normal values)
* Pregnancy
* Patients with treatment-resistant reflux symptoms. Defined as reflux persistent symptoms despite the use of a minimum dose of proton-pump inhibitors

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 130 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2023-05 (Actual)

PRIMARY OUTCOMES:
Percentage total body weight loss (%TBWL) | 3 years
  weight loss is measured in kilogram.

SECONDARY OUTCOMES:
Percentage excess weight loss (%EWL) | 3 years
  excess weight loss is measured in kilogram.
percentage total body weight regain (%TBWR) | 3 years
  Weight regain is measured in kilogram.
Decrease in type 2 diabetes mellitus | 3 years
  measuring glycated hemoglobin, decrease in diabetic medication
Quality of life | 3 years
  measuring BAROS score
Decrease in dyslipidaemia | 3 years
  decrease in medication for hypercholesterolaemie. Measuring cholesterol spectrum.
Decrease in hypertension | 3 years
  Measuring blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Rijnstate Hospital, Arnhem, Netherlands